CLINICAL TRIAL: NCT02442830
Title: A Comparison of Early Deployment of a Video Capsule (Endocapsule EC-10: Olympus Tokyo. Japan) in the Emergency Department Versus Standard of Care Workup of Non-hematemesis Gastrointestinal Bleeding
Brief Title: Comparing Early Capsule Deployment to Current Standard of Care for Management of Gastrointestinal Bleeding
Acronym: EDCAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Olympus Corporation (Industry)
Responsible Party: Principal Investigator, David Cave, Professor of Medicine, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H00006661
Record Dates: First submitted 2015-04-23; First posted 2015-05-13 (Estimated); Results first posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-07

CONDITIONS: Melena; Gastrointestinal Hemorrhage
MeSH Terms: conditions — Melena; Gastrointestinal Hemorrhage | interventions — Endoscopy; Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Early Video Capsule Endoscopy (Experimental): The intervention for subjects in this arm will be to have a video capsule deployed as soon as possible after presentation to the emergency department. Information from the video capsule will be obtained and reviewed to determine location of bleeding. Once that information has been obtained a decision will be made on which endoscopic test is most pertinent in finding and treating the source of bleeding.
  Interventions: Device: Early Video Capsule Endoscopy
- Standard of Care Workup Group (No Intervention): In this arm, patients will receive "standard of care workup" for non-hematemesis gastrointestinal bleeding. This could include upper endoscopy, colonoscopy, and additional capsule or small bowel enteroscopy depending on the subject's presentation and the results of the workup performed by the gastroenterology team. For patients requiring a video capsule endoscopy as part of "standard of care workup" the patients will be given the same Olympus video capsule that is used in the "Early Capsule" group.

INTERVENTIONS:
Device: Early Video Capsule Endoscopy — The intervention is the use of video capsule endoscopy as the first test in a patient presenting to the ED with active bleeding. The capsule allows for visualization of the entire GI tract.
  Once a capsule has been given to a study patient, a staff member will use the capsule's real-time viewer to see if there is any active bleeding in the stomach. If bleeding is seen the investigators will pursue an upper endoscopy. If no bleeding is seen a staff member will review the entire findings of the capsule and make a decision regarding which therapeutic measure to pursue.
  Other Names: Olympus Endocapsule 10 (EC-10) System
  Arms: Early Video Capsule Endoscopy

SUMMARY:
The objectives of this study are to test whether there are statistically significant differences between the standard of care workup workup of non-hematemesis gastrointestinal bleeding by endoscopy [upper, lower and other tests], compared with deployment of a video capsule as the first test followed by the most appropriate endoscopic procedure based on video capsule findings, if needed. The investigators propose to examine differences in time to diagnosis, reduction in numbers of procedures, and length of stay between a standard of care workup protocol and our proposed protocol of early capsule endoscopy deployment.

DETAILED DESCRIPTION:
After 40 years of considering gastrointestinal bleeding as upper or lower and largely ignoring the small intestine, there is accumulating evidence that the standard of care approach to the assessment of non-hematemesis gastrointestinal bleeding could be improved by early deployment of a video capsule (VCE) as the first diagnostic test. Currently, VCE is considered the gold standard as the diagnostic test for small intestinal bleeding. In a recent study at the University of Massachusetts (UMass) 336 patients who presented to the emergency department (ED) with complaints of gastrointestinal bleeding 36 patients (10.7%) were given a VCE during their stay.

In patients with hematemesis, upper endoscopy remains the diagnostic and therapeutic modality of choice. However patients with melena and hematochezia may benefit from early VCE since both signs and symptoms provide poor localization as to the origin of bleeding. Data from this previous Umass study suggests that the ingestion of a VCE in the ED could quickly and non-invasively provide clinicians accurate data as to the origin of the bleeding. This information could provide a guide to further management of the patient. VCE is able to visualize bleeding in the esophagus, stomach, duodenum, small intestine and right colon, thereby eliminating the guess work of deciding which endoscopic approach to use.

At UMass, that same study showed that of the 36 patients who received a video capsule, 26 (72.2%) had diagnostic studies (i.e. bleeding was identified). In comparison, 152 patients required upper endoscopy (of which 52.9% were diagnostic) and 64 patients required colonoscopy (of which 47% were diagnostic). Of those 26 patients with diagnostic capsule studies, 13 also required upper endoscopy, 1 required a colonoscopy, and 4 required both a colonoscopy and endoscopy. It is important to recognize, however, that often capsule studies are performed after upper endoscopy and colonoscopy and performed and are found to be negative. This sequence is the standard of care work up of bleeding. Despite being performed later in the hospital course of our patients, capsule studies have a high diagnostic yield. In reality VCE is used uncommonly in acute bleeding because it is rarely considered in the context of acute GI bleeding In this study, the investigators propose the approach of using the video capsule as the first diagnostic test prior to colonoscopy and endoscopy; this may lead to a shortened time to diagnosis, a reduction in length of stay, and a reduction in numbers of procedures due to early, accurate localization of the source of bleeding. All of these components could result in better quality of care and cost containment. Further, it is known that 80% of patients stop bleeding spontaneously. Thus the earlier they are examined the more likely the origin of the bleeding is likely to be found The use of VCE has been approved by the FDA since 2001 for small intestinal bleeding obscure GI Bleeding. It is very safe and no deaths associated with its use have been reported. More than two million capsules have been used and complications of obstruction and perforation are extremely rare.

Interest in the broader use of VCE is accumulating. More recently studies of VCE deployed in the ED, in patients with upper GI bleeding showed improved management. Our group recently demonstrated that the closer a VCE is performed to the time of bleeding the higher the likelihood of locating the sources and the higher the therapeutic intervention rate. The investigators also have demonstrated that the use of capsule endoscopy in patients with non-hematemesis gastrointestinal bleeding (NHGIB) has a higher diagnostic yield than does colonoscopy. With improved diagnostic yields, capsule endoscopy may help clinicians by providing guidance in the management of patients with NHGIB.

This protocol is be the first attempt to prospectively examine this concept in a large randomized prospective trial. The questions the investigators are studying are: can early capsule intervention decrease time to diagnosis, numbers of procedures and hospital length of stay in patients with non-hematemesis gastrointestinal bleeding?

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years old
* New onset of melena or hematochezia
* Able to sign consent
* Hemodynamically stable (i.e. blood pressure >100/60 or pulse <110 at the time of consent)
* ED must plan to admit patient to the hospital or Clinical Decision Unit.

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners
* Prior history of gastroparesis
* Prior history of gastric, or small bowel surgery
* Prior history of Crohn's disease
* Concern for infectious colitis
* Non-English speaking
* Evidence of dysphagia at the time of presentation
* Presence of bright red blood per rectum concerning for hemorrhoids
* Allergy to metoclopramide or erythromycin
* Code status of Do Not Resuscitate/Do Not Intubate (DNR/DNI) or Comfort Measures Only (CMO)
* Prior history of abdominal radiation
* Presence of Implantable Cardioverter Defibrillator (ICD) or pacemaker or other implanted electronic devices
* Abdominal pain suggesting an acute abdomen or obstruction. In clinical practice, only patients with crampy abdominal pain due to Crohn's disease, previous intestinal surgery and a previous history of radiation therapy require a patency capsule or CT enterography before capsule endoscopy.
* Patients who cannot undergo surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2015-04-19 (Actual); Primary Completion 2017-07-02 (Actual); Study Completion 2017-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Cave, MD, PhD, Principal Investigator — Professor of Medicine
Locations (1):
- University of Massachusetts Memorial Medical Center -- University Campus, Worcester, Massachusetts, United States

REFERENCES:
- [Background] Singh A, Marshall C, Chaudhuri B, Okoli C, Foley A, Person SD, Bhattacharya K, Cave DR. Timing of video capsule endoscopy relative to overt obscure GI bleeding: implications from a retrospective study. Gastrointest Endosc. 2013 May;77(5):761-6. doi: 10.1016/j.gie.2012.11.041. Epub 2013 Feb 1. PMID 23375526
- [Background] Jawaid S, Gondal B, Singh, A, Marshall C, and Cave D. The epidemiology of gastrointestinal bleeding in an academic emergency department as a basis for reconfiguring the conventional approach to its diagnosis and management. Gastrointestinal Endsocopy 2013;77:Supplement, Page AB483.
- [Background] Jawaid S, Marya N, Gondal B, Maranda L, Marshall C, Charpentier J, Singh A, Foley A, and Cave D. . A reconsideration of the diagnosis and management of gastrointestinal bleeding based on its epidemiology and outcomes analysis. Gastrointestinal Endsocopy 2014;79:Supplement, Page AB231.
- [Derived] Marya NB, Jawaid S, Foley A, Han S, Patel K, Maranda L, Kaufman D, Bhattacharya K, Marshall C, Tennyson J, Cave DR. A randomized controlled trial comparing efficacy of early video capsule endoscopy with standard of care in the approach to nonhematemesis GI bleeding (with videos). Gastrointest Endosc. 2019 Jan;89(1):33-43.e4. doi: 10.1016/j.gie.2018.06.016. Epub 2018 Jun 20. PMID 29935143

RESULTS

PARTICIPANT FLOW:
Groups:
- Early Video Capsule Endoscopy: The intervention for subjects in this arm will be to have a video capsule (VC) deployed as soon as possible after presentation to the emergency department. Information from the VC will be obtained and reviewed to determine location of bleeding. Once that information has been obtained a decision will be made on which endoscopic test is most pertinent in finding and treating the source of bleeding.
  Early VC Endoscopy (VCE): The intervention is the use of VCE as the first test in a patient presenting to the Emergency Department (ED) with active bleeding. The capsule allows for visualization of the entire bowel. Once a capsule has been given to a study patient, a staff member will use the capsule's real-time viewer to see if there is any active bleeding in the stomach. If bleeding is seen the investigators will pursue an upper endoscopy. If no bleeding is seen a staff member will review the entire findings of the VCE and make a decision regarding which therapeutic measure to pursue.
Period: Overall Study
Arm/Group | Early Video Capsule Endoscopy | Standard of Care Workup Group
Started | 42 | 45
Completed | 42 | 44
Not Completed | 0 | 1
Not completed — Technical Failure | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Early Video Capsule Endoscopy: The intervention for subjects in this arm will be to have a video capsule (VC) deployed as soon as possible after presentation to the emergency department. Information from the VC will be obtained and reviewed to determine location of bleeding. Once that information has been obtained a decision will be made on which endoscopic test is most pertinent in finding and treating the source of bleeding.
  Early Video Capsule Endoscopy: The intervention is the use of video capsule endoscopy as the first test in a patient presenting to the ED with active bleeding. The capsule allows for visualization of the entire GI tract.
  Once a capsule has been given to a study patient, a staff member will use the capsule's real-time viewer to see if there is any active bleeding in the stomach. If bleeding is seen the investigators will pursue an upper endoscopy. If no bleeding is seen a staff member will review the entire findings of the capsule and make a decision regarding which therapeutic me
- Total: Total of all reporting groups
Arm/Group | Early Video Capsule Endoscopy | Standard of Care Workup Group | Total
Number analyzed (Participants) | 42 | 45 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 13 | 34
  >=65 years | 21 | 32 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (12.6) | 70.4 (16.4) | 68.7 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 36
  Male | 23 | 28 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 39 | 43 | 82
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 36 | 42 | 78
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42 | 45 | 87
Type of bleeding at admission [Count of Participants; unit: Participants]
  Melena | 26 | 34 | 60
  Hematochezia | 11 | 9 | 20
  Symptomatic anemia | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Time to Localization of Bleeding
Description: Time to localization of bleeding refers to the time after a patient is admitted to the emergency room and a bleeding source is localized. We defined localization of bleeding as endoscopic visualization of stigmata of recent hemorrhage.
Time Frame: Enrollment to localization of bleeding as measured in hours, up to 720 hours, whichever is sooner.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Early Video Capsule Endoscopy | Standard of Care Workup Group
Number analyzed (Participants) | 42 | 45
hours | 21 [9 to 31] | 16 [13 to 31]
Statistical Analysis 1: Comparison: Early Video Capsule Endoscopy; Test type: Other — Log rank test; p = .002, Log Rank

2. Secondary Outcome: Number of Participants With Localization of Bleeding by the End of Admission
Description: This measurement counts the number of participants with a bleeding source localized by the end of admission.
Time Frame: Patient's will be assessed for the duration of their hospital stay and for thirty days afterwards.
Measure: Count of Participants; unit: Participants
Groups:
- Early Video Capsule Endoscopy: The intervention for subjects in this arm will be to have a video capsule (VC) deployed as soon as possible after presentation to the emergency department. Information from the VC will be obtained and reviewed to determine location of bleeding. Once that information has been obtained a decision will be made on which endoscopic test is most pertinent in finding and treating the source of bleeding.
  Early Video Capsule Endoscopy: The intervention is the use of VC endoscopy as the first test in a patient presenting to the ED with active bleeding. The capsule allows for visualization of the entire GI tract.
  Once a capsule has been given to a study patient, a staff member will use the capsule's real-time viewer to see if there is any active bleeding in the stomach. If bleeding is seen the investigators will pursue an upper endoscopy. If no bleeding is seen a staff member will review the entire findings of the capsule and make a decision regarding which therapeutic measure to pursue.
Arm/Group | Early Video Capsule Endoscopy | Standard of Care Workup Group
Number analyzed (Participants) | 42 | 45
Participants | 27 | 15

ADVERSE EVENTS:
Time Frame: 30 days
Description: Adverse events were collected only if they were considered procedure-related.
Groups:
- Early Video Capsule Endoscopy: The intervention for subjects in this arm will be to have a video capsule deployed as soon as possible after presentation to the emergency department. Information from the video capsule will be obtained and reviewed to determine location of bleeding. Once that information has been obtained a decision will be made on which endoscopic test is most pertinent in finding and treating the source of bleeding.
  Early Video Capsule Endoscopy: The intervention is the use of video capsule endoscopy as the first test in a patient presenting to the ED with active bleeding. The capsule allows for visualization of the entire GI tract.
  Once a capsule has been given to a study patient, a staff member will use the capsule's real-time viewer to see if there is any active bleeding in the stomach. If bleeding is seen the investigators will pursue an upper endoscopy. If no bleeding is seen a staff member will review the entire findings of the capsule and make a decision regarding which therapeutic me
Arm/Group | Early Video Capsule Endoscopy | Standard of Care Workup Group
All-Cause Mortality (participants affected / at risk) | 1/42 | 2/45
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/45
Other Adverse Events (participants affected / at risk) | 0/42 | 0/45

LIMITATIONS AND CAVEATS:
The study was performed in a single center with a relatively homogeneous population. Study personnel were not blinded to group allocation following randomization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-04-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT02442830/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT02442830/SAP_001.pdf